CLINICAL TRIAL: NCT04236726
Title: Investigating Health Related Quality of Life in Patients With Chronic Respiratory Failure
Acronym: CRF-QoL
Status: Recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CRF-QoL
Record Dates: First submitted 2019-12-17; First posted 2020-01-22 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Respiratory Failure; Neuromuscular Diseases; Ventilatory Failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency; Neuromuscular Diseases; Hypoventilation | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-invasive ventilation: Users of non-invasive ventilation
  Interventions: Other: Questionnaire
- Long term tracheostomy ventilation: Long term tracheostomy ventilated patients

INTERVENTIONS:
Other: Questionnaire — HRQoL questionnaires
  Groups: Non-invasive ventilation

SUMMARY:
To determine the quality of life of patients living with chronic respiratory failure and the impact interventions have on it.

DETAILED DESCRIPTION:
To determine the quality of life of patients living with chronic respiratory failure and the impact interventions have on it.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with chronic respiratory failure receiving any of:

* Non-invasive ventilation
* Prolonged mechanical ventilation
* Mechanical insufflation-exsufflation therapy

Exclusion Criteria:

* Aged <18
* Significant physical or psychiatric co-morbidity that would prevent compliance with trial protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic respiratory failure being treated with a form of ventilation of mechanical insufflation-exsufflation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-12-19 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
HRQoL score | Day 0: At the first outpatient clinical consultation with the clinical team
  Outcome of various HRQoL assessment tools.

SECONDARY OUTCOMES:
Change in HRQoL score | 6 months following first assessment for Outcome 1
  Change in HRQoL assessment tool score at next clinical follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Murphy, MBBS, Study Chair — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's and St. Thomas NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No